CLINICAL TRIAL: NCT00738699
Title: A Randomized, Double Blind, Placebo-Controlled Study of the Efficacy and Safety oF MORAb-003(Farletuzumab) in Combination With Paclitaxel Therapy in Subjects With Platinum-Resistant or Refractory Relapsed Ovarian Cancer
Brief Title: An Efficacy and Safety Study of MORAb-003 in Platinum-Resistant or Refractory Relapsed Ovarian Cancer
Acronym: FAR-122
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: study did not meet pre-specified criteria for continuation following interim futility analysis
Sponsor: Morphotek (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MORAb003-003PR
Record Dates: First submitted 2008-08-18; First posted 2008-08-20 (Estimated); Results first posted 2017-03-30 (Actual); Last update posted 2017-03-30 (Actual); Status verified 2017-02

CONDITIONS: Ovarian Cancer
Keywords: ovarian cancer; relapsed ovarian cancer; refractory ovarian cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — farletuzumab; Saline Solution; Paclitaxel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): MORAb-003 (Farletuzumab) Plus Paclitaxel
  Interventions: Drug: MORAb-003 (farletuzumab); Drug: Paclitaxel
- 2 (Placebo Comparator): Placebo Plus Paclitaxel
  Interventions: Drug: 0.9% Saline; Drug: Paclitaxel

INTERVENTIONS:
Drug: MORAb-003 (farletuzumab) — Farletuzumab (FAR) at 2.5 mg/kg was administered by intravenous (IV) infusion weekly on Day 1 of Weeks 1 to 12 (Cycle 1) and then in 4-week cycles with treatment administered on Day 1 of Weeks 1 to 3 for all subsequent cycles.
  Arms: 1
Drug: 0.9% Saline — Placebo (0.9% normal saline) was administered by IV infusion weekly on Day 1 of Weeks 1 to 12 (Cycle 1) and then in 4-week cycles with treatment administered on Day 1 of Weeks 1 to 3 for all subsequent cycles.
  Arms: 2
Drug: Paclitaxel
  Other Names: Paclitaxel (80 mg/m^2) was administered by IV infusion over 1 hour following administration of FAR.

SUMMARY:
The study is being conducted to find out if paclitaxel works better when given together with an experimental drug called MORAb-003 (farletuzumab) or alone in patients with platinum-resistant or refractory relapsed ovarian cancer

DETAILED DESCRIPTION:
Safety was assessed by the monitoring and recording of all adverse events (AEs), including drug hypersensitivity adverse events (DHAE), and serious adverse events (SAEs); clinical laboratory test (serum chemistry, hematology, urinalysis); tolerability (discontinuations, treatment delays, dose reductions); physical examinations (including vital signs assessment); 12-lead electrocardiograms (ECG) obtained in triplicate and reviewed by independent blinded cardiologist, and Karnofsky's performance status.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of non-mucinous epithelial ovarian cancer, including primary peritoneal and fallopian tube malignancies, measurable by CT or MRI scan assessed within 4 weeks prior to study entry
* Must have evidence of relapse by CA-125 (2xUpper Limit of Normal) or radiographically within 6 months of most recent platinum-containing chemotherapy. At least one of the lines of chemotherapy must have included a taxane.
* Must have been treated with debulking surgery and at least one line platinum-based chemotherapy;
* Subjects may have received up to four additional lines of chemotherapy after they developed platinum-resistance.
* Subjects must be candidate for repeat paclitaxel treatment

Exclusion Criteria:

* Clinical contraindications to use of paclitaxel, which include:

  1. persistent Grade 2 or greater peripheral neuropathy
  2. prior hypersensitivity reaction that persisted despite rechallenge with or without desensitization or resulted in bronchospasm or hemodynamic instability or was at least Grade 2 and resulted in medication discontinuation
* Current diagnosis of epithelial ovarian tumor of low malignant potential (borderline carcinomas). Note: EOC with prior diagnosis of a low malignant potential tumor that has been surgically resected is acceptable provided the subject did
* Prior radiation therapy is excluded with the exception that it is allowable only if measurable disease for ovarian cancer is completely outside the radiation portal
* Known allergic reaction to a prior monoclonal antibody therapy or have any documented human anti-human antibody (HAHA).
* Previous treatment with MORAb-003 (farletuzumab).

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 415 (Actual)
Dates: Start 2008-09; Primary Completion 2011-12 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (61):
- United States (34):
  - Southern Cancer Center, Mobile, Alabama
  - St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - California Cancer Care, Inc., Greenbrae, California
  - Moores UC San Diego Cancer Center, La Jolla, California
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Monterey Bay Oncology, Monterey, California
  - Jupiter Medical Center, Jupiter, Florida
  - Innovative Medical Research of South Florida, Inc., Miami, Florida
  - Florida Hospital Cancer Institute, Orlando, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - Memorial Health University Medical Center, Savannah, Georgia
  - Central DuPage Hospital, Winfield, Illinois
  - St. Vincent Gynecologic Oncology, Indianapolis, Indiana
  - Hematology and Oncology Specialists, LLC, Metairie, Louisiana
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Weinberg Cancer Institute at Franklin Square, Baltimore, Maryland
  - Henry Ford Health System, Detroit, Michigan
  - Morristown Memorial Hospital, Morristown, New Jersey
  - Schwartz Gynecologic Oncology, PLLC, Brightwaters, New York
  - Arena Oncology Associates, PC, Lake Success, New York
  - St. Luke's Roosevelt Hospital Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Piedmont Hematology Oncology Associates, PA, Winston-Salem, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Signal Point Clinical Research Center, Middletown, Ohio
  - Cancer Care Associates, Tulsa, Oklahoma
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Magee-Women's Hospital of UPMC, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - International Beneficence Clinical Research, LLC, Harlingen, Texas
  - South Texas Oncology & Hematology PA, San Antonio, Texas
  - Scott & White Memorial Hospital and Clinic, Temple, Texas
  - Utah Cancer Specialists, Salt Lake City, Utah
  - Northern Virginia Pelvic Surgery Associates, Annandale, Virginia
- Australia (9):
  - Prince of Wales Hospital, Randwick, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Royal Brisbane & Women's Hospital, Herston, Queensland
  - The Burnside War Memorial Hospital, Inc., Toorak Gardens, South Australia
  - Monash Medical Centre, East Bentleigh, Victoria
  - Mercy Hospital for Women, Heidelburg, Victoria
  - The Royal Women's Hospital, Parkville, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
  - St. John of God Hospital, Subiaco, Western Australia
- Belgium (3):
  - AZ Greninge Hospital, Kortrijk
  - University Hospitals Leuven, Leuven
  - CHU de Liege, Liège
- Canada (4):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - BC Cancer Agency, Kelowna, British Columbia
  - Juravinski Cancer Centre, Hamilton, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
- Netherlands (3):
  - UMCG, Groningen
  - University Hospital Maastricht, Maastricht
  - UMC Utrecht, Utrecht
- Spain (8):
  - Hospital Universitario Son Dureta, Palma de Mallorca, Balearic Islands
  - Hospital de Son Llatzer, Palma de Mallorca, Balearic Islands
  - Hospital Clinic I Provincial, Barcelona, Barcelona
  - Hospital de Mataro, Mataró, Barcelona
  - Corporacio Sanitaria Parc Taulis, Sabadell, Barcelona
  - Consorci Sanitari de Terrassa, Terrassa, Barcelona
  - Fundacion Hospital Alcorcon, Alcorcón, Madrid
  - Hospital Universitario 12 de Octubre, Madrid, Madrid

RESULTS

PARTICIPANT FLOW:
Groups:
- MORAb-003 (Farletuzumab) Plus Paclitaxel: Farletuzumab (FAR) at 2.5 mg/kg was administered by intravenous (IV) infusion weekly on Day 1 of Weeks 1 to 12 (Cycle 1) and then in 4-week cycles with treatment administered on Day 1 of Weeks 1 to 3 for all subsequent cycles. Paclitaxel (80 mg/m^2) was administered weekly by IV infusion over 1 hour following administration of FAR. During the 4-week cycle, Week 4 was to be a rest period with no study treatment (test article or paclitaxel) administered. All participants were required to be premedicated with steroids before paclitaxel administration, and with acetaminophen (650 mg orally) or clinically equivalent per clinic routine within 4 hours prior to test article infusion.
- Placebo (Normal Saline) Plus Paclitaxel: An equivalent volume of placebo (0.9% normal saline) was administered by IV infusion weekly on Day 1 of Weeks 1 to 12 (Cycle 1) and then in 4-week cycles with treatment administered on Day 1 of Weeks 1 to 3 for all subsequent cycles. Paclitaxel (80 mg/m^2) was administered weekly by IV infusion over 1 hour following administration of FAR. During the 4-week cycle, Week 4 was to be a rest period with no study treatment (test article or paclitaxel) administered. All participants were required to be premedicated with steroids before paclitaxel administration, and with acetaminophen (650 mg orally) or clinically equivalent per clinic routine within 4 hours prior to test article infusion.
Period: Overall Study
Arm/Group | MORAb-003 (Farletuzumab) Plus Paclitaxel | Placebo (Normal Saline) Plus Paclitaxel
Started | 275 | 140
Participants Not Treated | 2 | 1
Participants Treated | 273 | 139
Completed | 0 | 0
Not Completed | 275 | 140
Not completed — Withdrawal by Subject | 5 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Death | 144 | 68
Not completed — Discontinuation of study by Sponsor | 123 | 72
Not completed — Other | 2 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat population included, the primary population for the evaluation of efficacy, was defined as all participant who were randomly assigned to test article, analyzed by the treatment assigned.
Groups:
- Total: Total of all reporting groups
Arm/Group | MORAb-003 (Farletuzumab) Plus Paclitaxel | Placebo (Normal Saline) Plus Paclitaxel | Total
Number analyzed (Participants) | 275 | 140 | 415
Age, Continuous [Geometric Mean (Standard Deviation); unit: Years] | 60.9 (10.74) | 61.2 (9.44) | 61.0 (10.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 275 | 140 | 415
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: PFS was defined as the time (in months) from the date of randomization to the date of the first observation of progression as determined by modified Response Evaluation Criteria in Solid Tumors (RECIST), or death regardless of cause. If progression or death was not observed, the PFS time was censored at the date of the last tumor assessment without evidence of progression before the date of initiation of further antitumor treatment, or the cutoff date (whichever was earlier).
Time Frame: Date of Randomization to date of disease progression or death (whichever came first), assessed up to study termination (28 Nov 2011), or up to approximately 2 years 10 months
Population: Intent-To-Treat (ITT) population included all participants who were randomly assigned to study drug, analyzed by treatment assignment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | MORAb-003 (Farletuzumab) Plus Paclitaxel | Placebo (Normal Saline) Plus Paclitaxel
Number analyzed (Participants) | 275 | 140
Months | 3.5 [3.3 to 3.9] | 3.7 [3.3 to 5.2]
Statistical Analysis 1: Comparison: MORAb-003 (Farletuzumab) Plus Paclitaxel vs Placebo (Normal Saline) Plus Paclitaxel; Test type: Superiority or Other; p = 0.8360, Log Rank — One-sided log rank test stratified by route of administration for primary chemotherapy (intraperitoneal vs intravenous) and geographic region (North America, Europe, and other participating countries); Cox Proportional Hazard = 1.13, 95% CI 2-sided [0.88 to 1.46] — Stratified as described above

2. Primary Outcome: Overall Survival (OS)
Description: OS was defined as the time (in months) from the date of randomization to the date of death, whatever the cause. If death was not observed for a participant, the survival time was censored on the last date the participant was known to be alive or the cutoff date, whichever was earlier.
Time Frame: Date of Randomization to date of death, assessed up to study termination (28 Nov 2011), or up to approximately 2 years 10 months
Population: ITT population included all participants who were randomly assigned to study drug and analyzed by the treatment assigned.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | MORAb-003 (Farletuzumab) Plus Paclitaxel | Placebo (Normal Saline) Plus Paclitaxel
Number analyzed (Participants) | 275 | 140
Months | 11.3 [10.3 to 12.7] | 13.1 [10.3 to 16.7]
Statistical Analysis 1: Comparison: MORAb-003 (Farletuzumab) Plus Paclitaxel vs Placebo (Normal Saline) Plus Paclitaxel; Test type: Superiority or Other; p = 0.7568, Log Rank — One-sided log rank test stratified by route of administration for primary chemotherapy and geographic region; Cox Proportional Hazard = 1.11, 95% CI 2-sided [0.83 to 1.48] — Stratified as described above

3. Secondary Outcome: Best Overall Response
Description: BOR was defined as the percentage of participants having either a confirmed complete response (CR) or confirmed partial response (PR) using modified RECIST criteria by independent radiologist review. RECIST criteria was adjusted based on current medical practices and on possible differences between ovarian cancer and other solid tumors. Tumor assessments performed up to the initiation of further antitumor treatment were considered. Target lesions selected for response assessment were measured using computed tomography (CT) or magnetic resonance imaging (MRI) scans then graded according to the modified RECIST criteria, adjusted based on current medical practices and on possible differences between ovarian cancer and other solid tumors. Participants were assigned to one of the categories of change in disease state; CR, PR, progressive disease (PD), stable disease ( S)D, or not evaluable (NE).
Time Frame: Date of first study drug to disease progression/recurrence, assessed up to study termination (28 Nov 2011), or up to approximately 2 years 10 months
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | MORAb-003 (Farletuzumab) Plus Paclitaxel | Placebo (Normal Saline) Plus Paclitaxel
Number analyzed (Participants) | 275 | 140
Percentage of participants
  Complete response (CR) | 0.4 | 0
  Partial response (PR) | 7.3 | 15.0
Statistical Analysis 1: Comparison: MORAb-003 (Farletuzumab) Plus Paclitaxel vs Placebo (Normal Saline) Plus Paclitaxel; Test type: Superiority or Other; p = 0.0399, Cochran-Mantel-Haenszel — Compared the ratio of complete or partial responders in the two arms. Stratified by route of administration for first line therapy and geographic region as specified at baseline; Difference = -7.4, 95% CI 2-sided [-14.1 to -0.7] — (FAR + Paclitaxel) minus (Placebo + Paclitaxel). Confidence interval based on a normal approximation to the binomial distribution

4. Secondary Outcome: Time to Tumor Response (TTR)
Description: TTR was derived for those participants with objective evidence of CR or PR, and was defined as the time (in months) from the date of randomization to the first documentation of object tumor response (TR). Analysis was based on the Kaplan-Meier estimated percentage of responders. This statistical analysis method measures the effect of study drug on tumor response over a period of time.
Time Frame: Date of Randomization to the first documentation of objective TR, assessed up to study termination (28 Nov 2011), or up to approximately 2 years 10 months
Population: ITT population (Responders only) included all participants who were randomly assigned to study drug and analyzed by the treatment assigned.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | MORAb-003 (Farletuzumab) Plus Paclitaxel | Placebo (Normal Saline) Plus Paclitaxel
Number analyzed (Participants) | 21 | 21
Months | 2.0 [1.6 to 3.5] | 1.7 [1.6 to 3.3]

5. Other Pre Specified Outcome: Progression Free Survival Based on Gynecologic Cancer InterGroup (GCIG)
Description: Due to termination of the study, data were not collected and the outcome measure for PFS based on GCIG was not analyzed.
Time Frame: Length of study
Population: Due to termination of the study, data were not collected and the outcome measure for PFS based on GCIG was not analyzed.
Arm/Group | MORAb-003 (Farletuzumab) Plus Paclitaxel | Placebo (Normal Saline) Plus Paclitaxel
Number analyzed (Participants) | 0 | 0

6. Other Pre Specified Outcome: Serologic Response Rate
Description: Due to termination of the study, data were not collected and the outcome measure for Serologic Response Rate was not analyzed.
Time Frame: Length of study
Population: Due to termination of the study, data were not collected and the outcome measure for Serologic Response Rate was not analyzed.
Arm/Group | MORAb-003 (Farletuzumab) Plus Paclitaxel | Placebo (Normal Saline) Plus Paclitaxel
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: From the time the participant signed the study informed consent form until 30 days after the last dose of study drug (FAR or placebo), for up to approximately 3 years.
Description: Safety Analysis Set was defined as all randomized participants who received any dose of FAR or placebo, analyzed according to the test article received. The National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 3.0 was used to grade severity of AEs. Treatment-emergent adverse events were reported.
Arm/Group | MORAb-003 (Farletuzumab) Plus Paclitaxel | Placebo (Normal Saline) Plus Paclitaxel
Serious Adverse Events (participants affected / at risk) | 127/279 | 55/133
Other Adverse Events (participants affected / at risk) | 278/279 | 133/133
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MORAb-003 (Farletuzumab) Plus Paclitaxel (N=279) | Placebo (Normal Saline) Plus Paclitaxel (N=133)
Anaemia (Blood and lymphatic system disorders) | 7 | 7
Neutropenia (Blood and lymphatic system disorders) | 6 | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 4 | 1
Leukopenia (Blood and lymphatic system disorders) | 2 | 0
Atrial Fibrillation (Cardiac disorders) | 2 | 1
Cardiac Failure Congestive (Cardiac disorders) | 1 | 0
Cardio-Respiratory Arrest (Cardiac disorders) | 1 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 18 | 7
Intestinal Obstruction (Gastrointestinal disorders) | 10 | 4
Vomiting (Gastrointestinal disorders) | 9 | 5
Constipation (Gastrointestinal disorders) | 9 | 2
Ascites (Gastrointestinal disorders) | 8 | 2
Nausea (Gastrointestinal disorders) | 5 | 3
Abdominal Pain (Gastrointestinal disorders) | 5 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 3
Colonic Obstruction (Gastrointestinal disorders) | 3 | 0
Ileus (Gastrointestinal disorders) | 2 | 1
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 2 | 0
Gastrointestinal Obstruction (Gastrointestinal disorders) | 1 | 1
Intestinal Perforation (Gastrointestinal disorders) | 2 | 0
Large Intestinal Obstruction (Gastrointestinal disorders) | 1 | 1
Large Intestine Perforation (Gastrointestinal disorders) | 1 | 1
Abdominal adhesions (Gastrointestinal disorders) | 1 | 0
Colonic Pseudo-obstruction (Gastrointestinal disorders) | 1 | 0
Diverticulum (Gastrointestinal disorders) | 1 | 0
Enterocutaneous Fistula (Gastrointestinal disorders) | 1 | 0
Faecal Volume Decreased (Gastrointestinal disorders) | 1 | 0
Faecal Volume Increased (Gastrointestinal disorders) | 1 | 0
Gastric Ulcer (Gastrointestinal disorders) | 1 | 0
Gastrointestinal Inflammation (Gastrointestinal disorders) | 1 | 0
Gastrointestinal Perforation (Gastrointestinal disorders) | 1 | 0
Oesophageal Obstruction (Gastrointestinal disorders) | 1 | 0
Rectourethral Fistula (Gastrointestinal disorders) | 1 | 0
Short-Bowel Syndrome (Gastrointestinal disorders) | 1 | 0
Disease Progression (General disorders) | 17 | 7
Pyrexia (General disorders) | 15 | 2
Fatigue (General disorders) | 3 | 1
Asthenia (General disorders) | 1 | 1
Obstruction (General disorders) | 1 | 1
Pain (General disorders) | 1 | 1
Generalised Oedema (General disorders) | 1 | 0
Hernia Obstructive (General disorders) | 1 | 0
Oedema Peripheral (General disorders) | 1 | 0
Cholecystitis Acute (Hepatobiliary disorders) | 1 | 1
Cholangitis (Hepatobiliary disorders) | 1 | 0
Cellulitis (Infections and infestations) | 6 | 2
Urinary Tract Infection (Infections and infestations) | 5 | 3
Pneumonia (Infections and infestations) | 4 | 2
Sepsis (Infections and infestations) | 3 | 1
Catheter Site Infection (Infections and infestations) | 1 | 1
Device Related Infection (Infections and infestations) | 1 | 1
Infection (Infections and infestations) | 1 | 1
Lobar Pneumonia (Infections and infestations) | 1 | 1
Abdominal Infection (Infections and infestations) | 0 | 1
Bacterial Pyelonephritis (Infections and infestations) | 1 | 0
Candida Sepsis (Infections and infestations) | 1 | 0
Clostridium Difficle Colitis (Infections and infestations) | 1 | 0
Escherichia Sepsis (Infections and infestations) | 0 | 1
Herpes Zoster (Infections and infestations) | 1 | 0
Incision Site Infection (Infections and infestations) | 0 | 1
Infectious Peritonitis (Infections and infestations) | 0 | 1
Klebsiella Bacteraemia (Infections and infestations) | 0 | 1
Meningitis (Infections and infestations) | 0 | 1
Parotitis (Infections and infestations) | 1 | 0
Pelvic Infection (Infections and infestations) | 1 | 0
Postoperative Wound Infection (Infections and infestations) | 1 | 0
Pseudomonal Sepsis (Infections and infestations) | 1 | 0
Respiratory Tract Infection (Infections and infestations) | 1 | 0
Retroperitoneal Abcess (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 1 | 0
Postoperative Ileus (Injury, poisoning and procedural complications) | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0
Haemoglobin Decreased (Investigations) | 0 | 1
Weight decreased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 4 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 1 | 0
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Hypophagia (Metabolism and nutrition disorders) | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Fistula (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle Necrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Systemic Lupus Erythematosus (Musculoskeletal and connective tissue disorders) | 0 | 1
Oncologic Complication (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Metastases to Central Nervous System (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour Associated Fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Syncope (Nervous system disorders) | 2 | 1
Brain Mass (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 1 | 0
Encephelopathy (Nervous system disorders) | 0 | 1
Lethargy (Nervous system disorders) | 1 | 0
Mononeuritis (Nervous system disorders) | 0 | 1
Neuropathy Peripheral (Nervous system disorders) | 1 | 0
Posterior Reversible Encephelopathy Syndrome (Nervous system disorders) | 1 | 0
Depression (Psychiatric disorders) | 2 | 1
Anxiety (Psychiatric disorders) | 1 | 0
Disorientation (Psychiatric disorders) | 1 | 0
Mental Status Change (Psychiatric disorders) | 1 | 0
Renal Failure Acute (Renal and urinary disorders) | 2 | 2
Hydronephrosis (Renal and urinary disorders) | 2 | 1
Renal Failure (Renal and urinary disorders) | 1 | 2
Bladder Spasm (Renal and urinary disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 1 | 0
Renal Impairment (Renal and urinary disorders) | 0 | 1
Ureteric Obstruction (Renal and urinary disorders) | 1 | 0
Urinary Tract Obstruction (Renal and urinary disorders) | 1 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 10 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 | 4
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 5 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dermatits Exfoliative (Skin and subcutaneous tissue disorders) | 0 | 1
Palmar-Plantar Erythrodysaesthesia Syndrome (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Skin Toxicity (Skin and subcutaneous tissue disorders) | 1 | 0
Hypotension (Vascular disorders) | 2 | 2
Thrombosis (Vascular disorders) | 3 | 0
Deep Vein Thrombosis (Vascular disorders) | 1 | 1
Subclavian Vein Thrombosis (Vascular disorders) | 1 | 0
Superior Vena Cava Syndrome (Vascular disorders) | 0 | 1
Venous Thrombosis Limb (Vascular disorders) | 1 | 0
Pneumonia bacterial (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MORAb-003 (Farletuzumab) Plus Paclitaxel (N=279) | Placebo (Normal Saline) Plus Paclitaxel (N=133)
Nausea (Gastrointestinal disorders) | 132 | 66
Diarrhoea (Gastrointestinal disorders) | 119 | 53
Constipation (Gastrointestinal disorders) | 96 | 53
Abdominal pain (Gastrointestinal disorders) | 88 | 34
Vomiting (Gastrointestinal disorders) | 84 | 37
Abdominal Distension (Gastrointestinal disorders) | 51 | 21
Ascites (Gastrointestinal disorders) | 22 | 11
Stomatitis (Gastrointestinal disorders) | 26 | 7
Dyspepsia (Gastrointestinal disorders) | 22 | 10
Abdominal Pain Upper (Gastrointestinal disorders) | 25 | 6
Dry mouth (Gastrointestinal disorders) | 19 | 8
Small intestinal Obstruction (Gastrointestinal disorders) | 19 | 7
Flatulence (Gastrointestinal disorders) | 18 | 5
Gastroresophageal Reflux Disease (Gastrointestinal disorders) | 10 | 8
Fatigue (General disorders) | 184 | 82
Oedema Peripheral (General disorders) | 60 | 26
Pyrexia (General disorders) | 43 | 18
Asthenia (General disorders) | 24 | 12
Mucosal Inflammation (General disorders) | 24 | 11
Chills (General disorders) | 18 | 7
Disease Progression (General disorders) | 17 | 7
Pain (General disorders) | 17 | 7
Oedema (General disorders) | 6 | 7
Neuropathy Peripheral (Nervous system disorders) | 75 | 37
Headache (Nervous system disorders) | 72 | 28
Dizziness (Nervous system disorders) | 42 | 18
Peripheral Sensory Neuropathy (Nervous system disorders) | 38 | 15
Dysguesia (Nervous system disorders) | 29 | 22
Restless Legs Syndrome (Nervous system disorders) | 14 | 2
Hypoaesthesia (Nervous system disorders) | 6 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 58 | 27
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 56 | 21
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 50 | 25
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 29 | 6
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 16 | 13
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 9 | 9
Urinary Tract Infection (Infections and infestations) | 47 | 30
Upper Respiratory Tract Infection (Infections and infestations) | 24 | 6
Nasopharyngitits (Infections and infestations) | 16 | 4
Sinusitis (Infections and infestations) | 10 | 9
Arthralgia (Musculoskeletal and connective tissue disorders) | 43 | 22
Back Pain (Musculoskeletal and connective tissue disorders) | 36 | 26
Myalgia (Musculoskeletal and connective tissue disorders) | 28 | 17
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 31 | 12
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 14 | 12
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 15 | 6
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 14 | 6
Decreased Appetite (Metabolism and nutrition disorders) | 67 | 27
Hypomagnesaemia (Metabolism and nutrition disorders) | 31 | 18
Hypokalaemia (Metabolism and nutrition disorders) | 28 | 9
Dehydration (Metabolism and nutrition disorders) | 14 | 5
Anaemia (Blood and lymphatic system disorders) | 78 | 37
Neutropenia (Blood and lymphatic system disorders) | 38 | 18
Leukopenia (Blood and lymphatic system disorders) | 16 | 9
Insomnia (Psychiatric disorders) | 54 | 23
Anxiety (Psychiatric disorders) | 25 | 16
Depression (Psychiatric disorders) | 24 | 8
Flushing (Vascular disorders) | 28 | 9
Hypotension (Vascular disorders) | 10 | 7
Dysuria (Renal and urinary disorders) | 9 | 12
Pollakiuria (Renal and urinary disorders) | 7 | 9
Contusion (Injury, poisoning and procedural complications) | 19 | 1
Vision Blurred (Eye disorders) | 14 | 8
Alopecia (Skin and subcutaneous tissue disorders) | 143 | 59
Rash (Skin and subcutaneous tissue disorders) | 55 | 19
Nail disorder (Skin and subcutaneous tissue disorders) | 47 | 19
Dry skin (Skin and subcutaneous tissue disorders) | 18 | 7
Erythema (Skin and subcutaneous tissue disorders) | 18 | 6
Pruritus (Skin and subcutaneous tissue disorders) | 15 | 8
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 13 | 7
Nail discolouration (Skin and subcutaneous tissue disorders) | 11 | 7

LIMITATIONS AND CAVEATS:
This study was prematurely terminated by the sponsor following results of the preplanned futility analysis showing the study was unlikely to meet its statistically-defined coprimary endpoints.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other